CLINICAL TRIAL: NCT00004430
Title: Randomized Study of Photodynamic Therapy Using Dihematoporphyrin in Patients With Corneal Neovascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Hampton Roads (Other)
Collaborators: Eastern Virginia Medical School (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13380; EVMS-FDR001020
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-08

CONDITIONS: Corneal Neovascularization
Keywords: cardiovascular and respiratory diseases; corneal neovascularization; rare disease
MeSH Terms: conditions — Corneal Neovascularization; Respiratory Tract Diseases; Rare Diseases | interventions — Prednisolone; Laser Therapy

INTERVENTIONS:
Drug: Dihematoporphyrin derivative
Drug: prednisolone
Procedure: Laser surgery

SUMMARY:
OBJECTIVES:

I. Demonstrate the safety and efficacy of dihematoporphyrin derivative (DHP) in laser photodynamic therapy (PDT) in patients with corneal neovascularization.

II. Document the histopathologic mechanism of action in selected patients undergoing penetrating keratoplasty following PDT therapy for corneal neovascularization.

III. Facilitate FDA product approval of DHP as a photosensitizing agent for laser treatment in these patients.

IV. Explore the use of this photosensitizer for ocular and cutaneous basal cell and squamous cell carcinoma.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, placebo controlled study.

Patients are randomized to 1 of 3 treatment arms:

Arm I: Patients receive topical dihematoporphyrin derivative (DHP) every 3 hours on days -3 and -2. Patients undergo laser surgery on day 0. After photodynamic (PDT) therapy, patients receive topical prednisolone phosphate four times a day for 90 days. Ninety days following PDT, patients may undergo corneal transplantation.

Arm II: Patients receive placebo topical gel and undergo sham laser surgery following arm I schedule, then receive topical prednisolone phosphate four times a day for 90 days. Patients may be crossed over to arm I if disease progression is observed.

Arm III: Patients receive a compressed 1 day schedule of DHP with 5 doses in the morning and then undergo laser surgery in the evening.

Patients are assessed on days 1, 7, 30, and 90 after PDT therapy.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
* Histologically proven corneal neovascularization (CNV): Must have at least 1 quadrant of significant CNV, which is due to bacterial, viral, parasitic, or fungal keratitis; alkaline acid or hydrocarbon chemical burns; ocular trauma and injury; severe ocular surface disease; or previous surgery with complications such as corneal allograft rejection are eligible
* No concurrent systemic steroids
* No concurrent immunosuppressive therapy
* Not pregnant or nursing; Negative pregnancy test; Fertile patients must use effective contraception; HIV negative; No rheumatoid arthritis; No congenital corneal scars; No active ocular infection or inflammation; No other active systemic collagen vascular disease; No uncontrolled glaucoma; No history of porphyrin allergies; Visual acuity of 20/400 or better in contralateral eye

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 1994-09; Study Completion 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: John D. Sheppard, Study Chair — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

REFERENCES:
- [Background] Sheppard JD, Chames MA, Clarke KC, et al.: Argon laser photodynamic thrombosis of human corneal neovascularization utilizing intravenous dihematoporphyrin. Investigative Ophthalmology and Visual Science 35(4): 1350, 1994.
- [Background] Chames MA, Sheppard JD, Mittal DC, et al.: A rabbit model for argon laser photodynamic therapy of corneal neovascularization utilizing topical dihematoporphyrin. Investigative Ophthalmology and Visual Science 36(1): 146, 1995.
- [Background] Mittal DC, Chames MS, Sheppard JD, et al.: Distribution of dihematoporphyrin in rabbit cornea, iris, aqueous humor and plasma after topical intravenous administration. Investigative Ophthalmology and Visual Science 36(13): 2564, 1995.
- [Background] Lattanzio F, Rusch A, Sheppard J, et al.: Documentation of corneal neovascularization by quantitative video fluorescein angiography. Investigative Ophthalmology and Visual Science 37: S546, 1996.
- [Background] Cox KW, Sheppard JD, Lattanzio FA, et al.: Photodynamic therapy of corneal neovascularization using topical dihematoporphyrin ester. Investigative Ophthalmology and Visual Science 38: S512, 1997.
- [Background] Williams PB, Sheppard JD, Chames MA, et al.: Distribution of dihematoporphyrin in rabbit cornea, iris, aqueous humor and serum after topical vs intravenous administration. Journal of Clinical Pharmacology 35(10): 936, 1995.